CLINICAL TRIAL: NCT03778970
Title: Pain Neuroscience Education vs. Self-management Programs Associated With Movement Control Exercises for Chronic Low Back Pain: a Randomized Controlled Clinical Study
Brief Title: Pain Education vs. Self-management Associated With Movement Control Exercises for Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Thais Cristina Chaves, Professor PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69172017.1.0000.5440
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial, superiority trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will be submitted to Pain Neuroscience Education or Self-Management Education plus movement control exercises. They will not be aware of the education approach they will receive. The assessors will also not be aware whether the participant received Pain Neuroscience Education or Self-Management Education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education + Exercises (Experimental): The PNE will follow the principles established by Explain Pain, addressing reconceptualization of pain, emphasizing modern neuroscience concepts. The PNE workshop will last 40 minutes (2 sessions). The movement control exercises will consist of active exercises that address posture and control of movements which are impaired and trigger pain. The session will last approximately 30 minutes, starting with the execution of the coordination exercises in the control of movement with an intensity of 10 to 30 repetitions and then performing exercises for stretching in 3 series of 30 seconds. Finally, strengthening exercises in 3 sets of 15 repetitions will be implemented. The exercises will be administered 1 session/week (volunteers will be oriented to execute the same exercises at home twice a week). The volunteers will receive 8 sessions at the clinic.
  Interventions: Other: Pain Neuroscience Education; Other: Movement Control Exercises
- Self-Management Education + Exercises (Active Comparator): The Self-Management Education (SME) strategy will be aligned with the "Back Book" concepts, focused on behavior change and encouraging participants to be active despite of the pain. The SME workshop will last 40 minutes (2 sessions). The movement control exercises will consist of active exercises that address posture and control of movements which are impaired and trigger pain. The session will last approximately 30 minutes, starting with the execution of the coordination exercises in the control of movement with an intensity of 10 to 30 repetitions and then performing exercises for stretching in 3 series of 30 seconds. Finally, strengthening exercises in 3 sets of 15 repetitions will be implemented. The exercises will be administered 1 session/week (volunteers will be oriented to execute the same exercises at home twice a week). The volunteers will receive 8 sessions at the clinic.
  Interventions: Other: Self-Management Education; Other: Movement Control Exercises

INTERVENTIONS:
Other: Pain Neuroscience Education — Pain neuroscience education (2 sessions during 40 minutes) administered by an interactive workshop
  Arms: Pain Neuroscience Education + Exercises
Other: Self-Management Education — A self-management education (2 sessions during 40 minutes) administered by an interactive workshop
  Arms: Self-Management Education + Exercises
Other: Movement Control Exercises — Eight sessions of movement control exercises (30 minutes each) + advice to perform the exercises at home twice a week.

SUMMARY:
The primary aim of this study is to compare the effects of an exercise program based on movement control exercises associated with self-management advice (SME) or pain neuroscience education (PNE) on the outcomes of pain intensity and pain disability in patients with chronic non-specific low back pain (CLBP).

DETAILED DESCRIPTION:
Participants: One hundred and four volunteers (104) aged 18-50 years with chronic non-specific low back pain.

Interventions: The volunteers will be randomized into two treatment groups: self-management education and movement control exercises or pain neuroscience education and exercises based on movement control exercises. Two workshops of 40 minutes each will be administered as education approach and the exercise program along 2 months ( and 12 sessions distributed over 2 months.

Main outcome measures: Primary outcomes will include pain intensity and low back disability, and secondary outcomes will be pain catastrophizing, pain self-efficacy, kinesiophobia, exercise adherence and global perceived effect. These will be measured pre- and post-intervention and at the 1-month follow-up. Statistical analysis will be conducted following treatment intent principles, and treatment effects will be calculated using a mixed linear model, considering intervention groups as a factor and assessments over time as repeated measures.

ELIGIBILITY:
Inclusion Criteria:

(1) non-specific chronic low back pain with a mechanical constituent caused by certain postures, activities, and movements, in addition to having at least 3 months of pain and/or episodes for at least half the previous 6 days, located between T12 and the gluteal folds; (2) pain intensity scores greater than 2 and greater than 14% on the Oswestry Low Back Disability Index and (3) positive results in 2 or more of the 6 tests to determine movement control impairment.

Exclusion Criteria:

(1) red flags such as tumors or neoplastic diseases in the spine, inflammatory diseases, infections, and fractures; (2) central and peripheral, psychiatric, rheumatologic, and cardiac neurological diseases; (3) acute and symptomatic radiculopathy, lumbar stenosis, and spondylolisthesis; (4) pregnant women; and (5) individuals submitted to physiotherapeutic treatment during the last 6 months. Finally, volunteers will be advised about the non-use of pain medications 24 hours before the evaluations.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity - Numerical Pain Rating Scale (NPRS) | Immediately after and at 1-month follow-up
  The NPRS used to assess pain intensity in this trial will consist in a sequence of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable". Previous research has found the NPRS to be responsive to change, with a minimum clinically important difference (MCID) of 2.4 among patients with CLBP receiving exercise or education.
Low Back Pain Disability | Immediately after and at 1-month follow-up
  The Brazilian Portuguese version of Oswestry Disability Index (ODI) will be used to assess low back pain related disability. This instrument consists of 10 items, each of which has six response options. The total score will be calculated by summing up all the points, with the largest possible sum being 50. This sum will be transformed into a percentage by multiplying it by two. Previous research has found that ODI showed responsiveness to change for patients with CLBP, with MCID of 8 points.

SECONDARY OUTCOMES:
Pain Catastrophizing | Immediately after and at 1-month follow-up
  Validated and translated to Brazilian-Portuguese, the Pain Catastrophizing scale (Br-PCS) is a self-administered questionnaire that presents 13 questions, divided into 3 domains: helplessness, magnification, and rumination. The scale has 5 points: 0 (minimum); 1 (slight); 2 (moderate); 3 (intense); and 4 (very intense). The final score ranges from 0 to 52 points, with the psychological risk being directly proportional to higher scores.
Pain Self-Efficacy | Immediately after and at 1-month follow-up
  Validated for Brazilian-Portuguese, the Pain Self-Efficacy Scale (PSE) presents 10 questions scored from 0 (Not at all confident) to 6 (Completely confident). The score achieved on this scale can range from 0 to 60, higher values reflecting stronger self-efficacy beliefs.
Fear Avoidance Beliefs | Immediately after and at 1-month follow-up
  Validated and translated to Brazilian-Portuguese, the Fear Avoidance Beliefs Questionnaire (FABQ-Brazil) is composed of 16 self-report items, subdivided into the FABQ-Phys, addressing beliefs related to occupational activities, and the FABQ-Work, work-related beliefs. However, the FABQ-Work score should be measured by adding items 6,7,9,10,11,12, and 15 with a score ranging from 0 to 42 and the FABQ-Phys through the sum of items 2,3,4, and 5, with the score ranging from 0 to 24 points.
Exercise Adherence | at the beginning of following session, immediately after and at 1-month follow-up
  We will administer the Brazilian Portuguese version of the scale cross-culturally adapted. The tool is comprised of 16 items, 6 items directly assessing behavior adherence (Section B), while 10 additional items related to non-adherence reasons (Section C). The 16 items were classified using an ordinal scale of 5 possible answers (0 = strongly agree to 4 = totally disagree) with a possible score range from 0 to 64. A higher overall adherence score indicated better adherence to exercise.
Global Perceived Effect | Immediately after and at 1-month follow-up
  The Global Perceived Effect Scale has the purpose of investigating musculoskeletal features, where the patient has the capacity to report improvement or deterioration over time, usually used to measure the effect of a therapy with the question: "Compared to when this episode began, how would you describe your low back currently?" Scored from -5 (much worse) to +5 (fully recovered), higher scores indicate improvement in the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Thais Chaves, PhD, Study Director — Professor - Ribeirão Preto Medical School - University of São Paulo
Locations (2):
- Brazil (2):
  - Physical Therapy Clinic, Jacarezinho, Paraná
  - University of Sao Paulo, Ribeirão Preto, São Paulo